CLINICAL TRIAL: NCT01391533
Title: Dose Escalation, Safety, Pharmacokinetic and Pharmacodynamic, First in Man Study, of SAR125844 Single Agent Administered as Slow Intravenous Infusion in Adult Patients With Advanced Malignant Solid Tumors
Brief Title: Study of SAR125844 Single Agent Administered as Slow Intravenous Infusion in Adult Patients With Advanced Malignant Solid Tumors
Acronym: SARMET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TED11449; 2010-021398-36 (EudraCT Number); U1111-1117-9878 (Other: UTN)
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Malignant Solid Tumors
MeSH Terms: interventions — SAR125844

ARMS (1):
- Dose Escalation (Experimental): Dose escalation phase: The starting dose of SAR125844 will be 50 mg/m^2 up to 960 mg/m^2
  Interventions: Drug: SAR125844

INTERVENTIONS:
Drug: SAR125844 — Pharmaceutical form:solution
  Route of administration: intravenous

SUMMARY:
Primary Objectives:

To determine the maximum tolerated dose (MTD) of SAR125844. To confirm safety profile of SAR125844 when administered as single agent at the MTD.

To evaluate the preliminary anti-tumoral effect of SAR125844 in patients with MET-gene amplified solid tumors (including sub-group of MET-amplified non-small cell lung cancer [NSCLC] patients) and in patients with Phospho-MET positive tumors without MET-gene amplification.

Secondary Objectives:

To characterize the global safety profile including cumulative toxicities. To evaluate the pharmacokinetic profile of SAR125844 in the proposed dosing schedule(s).

To assess preliminary antitumor activity in patients with measurable/evaluable disease, according to RECIST 1.1 criteria.

To explore the pharmacodynamic effects (PD) of SAR125844. To explore MET gene amplification status in Circulating Tumoral Cells (CTCs) and on tumor biopsies collected during the study, in the escalation part only.

To evaluate other pharmacodynamic biomarkers and help selection of patients who could benefit from SAR125844.

To explore MET-gene amplification status in circulating DNA.

DETAILED DESCRIPTION:
The duration of the study for one patient in the dose escalation phase of the study will include a screening period of up to 3 weeks and a 4-week treatment cycle(s). The patients may continue treatment until disease progression, unacceptable toxicity, or willingness to stop, followed by a minimum of 30-day follow-up. The study will also include 2 expansion cohorts. If a patient treated in dose escalation part or in an expansion cohorts, continues to benefit from the treatment at the time of Clinical Study Report, the patient can continue study treatment for a maximum of 1 year and will continue to undergo all assessments as per the study flowchart. Such patients will be followed at least until 30 days after the last IMP administration.

ELIGIBILITY:
Inclusion criteria:

In the dose escalation part: patients with high MET tumor expression, evaluable or measurable solid tumors for which no standard therapy is available.

In the expansion cohorts: in the first cohort, patients with diagnosed MET gene amplified including NSCLC patients and measurable tumors for which no standard therapy is available will be eligible. In the second cohort, patients with advanced P-MET positive measurable solid tumor without MET- gene amplification for which no standard therapy is available will be eligible.

Exclusion criteria:

Patient less than 18 years old. ECOG performance status >2. Any serious active disease or co-morbid condition, which, in the opinion of the Investigator, may interfere with the safety or the compliance with the study.

Poor bone marrow reserve as defined by absolute neutrophil count <1.5 x 10^9/L or platelets <100 x 10^9/L.

Poor organ function as defined by one of the following:

* Total bilirubin >1.5 x ULN
* AST, ALT, alkaline phosphatase >2.5 x ULN or >5 x ULN in case of documented liver metastasis. Alkaline phosphatase up to 5 x ULN in case of osteolytic bone metastasis without liver metastases is allowed
* Serum creatinine >1.5 x ULN or
* Serum creatinine between 1.0 and 1.5 x ULN associated with calculated creatinine clearance <60 mL/min
* Proteinuria >500 mg/24H Pregnant or breast-feeding women. No use of effective birth control methods, when applicable. No measurable or evaluable tumor lesion in the Dose Escalation part, and no measurable lesions in the expansion cohorts.

Brain metastasis (other than totally resected or previously pre-irradiated and no progressive/relapsing) or lepto-meningeal carcinomatosis.

No resolution of any specific toxicities (excluding alopecia) related to any prior anti-cancer therapy to grade ≤1 according to the NCI CTCAE v.4.03.

Wash out period of less than 3 weeks from previous antitumor therapy or any investigational treatment (and less than 6 weeks in case of prior nitroso-urea and or mitomycin C treatment).

Any surgery with major risk of bleeding performed less than 10 days prior to study treatment administration.

Any other severe underlying medical conditions, which could impair the ability to participate in the study or the interpretation of its results.

Patients treated with potent CYP3A inhibitor unless it can be discontinued at least 2 weeks prior to study treatment or 5 elimination half-life, whichever is the longest.

Patients treated with potent and moderate CYP3A inducers unless it can be discontinued at least 2 weeks prior to study treatment or 5 elimination half-life, whichever is the longest. Patients treated with weak CYP3A inducers such as dexamethasone are eligible.

Known hypersensitivity or any adverse event related to the study drug excipient.

Prior treatment with any compound in the same class. Mean QTc interval prolongation.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Dose Escalation To determine the maximum tolerated dose (MTD) of SAR125844 | At day 28 of Cycle 1 of each treated patient, DLT is assessed
Expansion Cohorts To evaluate the preliminary anti-tumoral effect of SAR125844 | Anticancer activity is assessed at Day 28 and then every 8 weeks thereafter up to an expected maximum of 2 years

SECONDARY OUTCOMES:
Number of patients with treatment emergent events | Up to 2 years
Assessment of PK parameter Cmax | Up to 2 years
Assessment of PK parameter AUCs | Up to 2 years
Assessment of PK parameter CL | Up to 2 years
Assessment of PD parameter ShedMET | Up to 2 years
Assessment of PD parameter HGF | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Investigational Site Number 840001, Boston, Massachusetts, United States
- France (2):
  - Investigational Site Number 250002, Dijon
  - Investigational Site Number 250001, Villejuif
- Italy (3):
  - Investigational Site Number 380004, Bologna
  - Investigational Site Number 380002, Milan
  - Investigational Site Number 380001, Milan
- Spain (2):
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724003, Madrid

REFERENCES:
- [Derived] Angevin E, Spitaleri G, Rodon J, Dotti K, Isambert N, Salvagni S, Moreno V, Assadourian S, Gomez C, Harnois M, Hollebecque A, Azaro A, Hervieu A, Rihawi K, De Marinis F. A first-in-human phase I study of SAR125844, a selective MET tyrosine kinase inhibitor, in patients with advanced solid tumours with MET amplification. Eur J Cancer. 2017 Dec;87:131-139. doi: 10.1016/j.ejca.2017.10.016. Epub 2017 Nov 14. PMID 29145039